CLINICAL TRIAL: NCT06973031
Title: A Prospective Clinical Study to Evaluate the Safety and Effectiveness of Pulmonary Vein Isolation Plus Box Isolation of Fibrotic Areas With the Globe® Pulsed Field System for Treating Patients With Symptomatic Paroxysmal or Persistent Atrial Fibrillation
Acronym: GLOBAL-PF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kardium Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-285345
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-06-16 (Actual); Status verified 2025-06

CONDITIONS: Paroxysmal Atrial Fibrillation (PAF); Persistent Atrial Fibrillation
Keywords: Pulsed Field Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Globe Pulsed Field System (Experimental)
  Interventions: Device: Globe Pulsed Field System

INTERVENTIONS:
Device: Globe Pulsed Field System — Ablation and atrial mapping with the Globe Pulsed Field System

SUMMARY:
The study will evaluate the safety and 12-month effectiveness of the Pulmonary Vein Isolation plus Box Isolation of Fibrotic Areas (BIFA) ablation strategy with the Globe Pulsed Field System (Globe PF System) for the treatment of atrial fibrillation.

ELIGIBILITY:
Key inclusion criteria:

* A diagnosis of recurrent symptomatic paroxysmal or persistent AF
* Failure or intolerance of at least one antiarrhythmic drug (AAD) Class I or III

Key exclusion criteria:

* Long-standing persistent AF (sustained >12 months)
* Atrial fibrillation secondary to a reversible cause or of non-cardiac origin
* History of thromboembolic events within the past six months
* Myocardial infarction (MI)/percutaneous coronary intervention (PCI) within the last three months
* Any cardiac surgery within the previous six months
* Prior left atrial ablation or surgical procedure
* Presence of an implanted cardiac device
* Body mass index (BMI) >40 kg/m^2
* Left ventricular ejection fraction (LVEF) <35%
* Anterior-posterior left atrial (LA) diameter >55mm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness endpoint | 12 months
  Number of subjects with freedom from documented atrial fibrillation, atrial flutter, and atrial tachycardia (AF/AFL/AT) 12 months post-procedure.
Safety endpoint | 7 days
  Rate of subjects presenting with one or more of the specified primary safety events within 7 days of the index ablation procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Westpfalz-Klinikum GmbH Kaiserslautern, Kaiserslautern, Germany